CLINICAL TRIAL: NCT01888172
Title: Weight Watchers Online
Acronym: WWO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: WW International Inc (Industry); University of Tennessee (Other)
Responsible Party: Principal Investigator, John Graham Thomas, Assistant Professor (Research), The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WeightWatchersOnline
Record Dates: First submitted 2013-06-24; First posted 2013-06-27 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Eating

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Weight Watchers Online (Experimental)
  Interventions: Behavioral: Weight Watchers Online Program
- Weight Watchers Online + ActiveLink (Experimental)
  Interventions: Behavioral: Weight Watchers Online Program; Device: Philips ActiveLink
- Internet Delivered Eating and Activity Program (Active Comparator)
  Interventions: Behavioral: Eating and Activity Newsletter

INTERVENTIONS:
Behavioral: Weight Watchers Online Program — Access to the Weight Watchers Online program available via the Internet on personal computers, tablet computers, and smartphones.
  Arms: Weight Watchers Online; Weight Watchers Online + ActiveLink
Device: Philips ActiveLink — Provision of a key-chain sized physical activity monitor that interfaces with the Weight Watchers website to promote exercise and give feedback on progress towards exercise goals.
  Arms: Weight Watchers Online + ActiveLink
Behavioral: Eating and Activity Newsletter — General information on healthy eating and physical activity habits and the medical consequences of overweight/obesity and weight loss.
  Arms: Internet Delivered Eating and Activity Program

SUMMARY:
The purpose of this study is to conduct a randomized controlled trial to compare the weight losses produced by the Weight Watchers Online program (WWO) and WWO plus the Philips ActiveLink physical activity system, over a 1-year period, compared to a control group.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 27 and 40 kg/m2
* All ethnic groups will be recruited
* English speaking
* Have access to the Internet via a computer, and basic computer skills

Exclusion Criteria:

* Report health problems that make weight loss or unsupervised exercise unsafe or unreasonable
* Report a heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire
* Are currently pregnant or breastfeeding, or intend to become pregnant in the next 12 months
* Are planning to move outside of the state within the next 12 months
* Report any cognitive or physical limitations that preclude use of a personal computer
* Have participated in a study conducted by the WCDRC or UT in the past 2 years
* Have followed a commercial weight-loss program within the previous 6 months or who are currently following a commercial weight loss program
* Weight loss of ≥ 5% of initial body weight in the last 6 months
* History of clinically diagnosed eating disorder excluding Binge Eating Disorder.
* Previous surgical procedure for weight loss
* Currently taking weight loss medication
* Treatment of cancer within the last 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in body weight, measured in kilograms | 3, 6, 9, and 12 months after randomizaiton

SECONDARY OUTCOMES:
Engagement with the electronic intervention system | 3, 6, 9, and 12 months after randomization
  The frequency with with participants interact with the Weight Watchers Online and control group websites.
Blood pressure | 3, 6, 9, and 12 months after randomization

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Miriam Hospital Weight Control & Diabetes Research Center, Providence, Rhode Island
  - University of Tennessee, Knoxville, Tennessee

REFERENCES:
- [Derived] Thomas JG, Raynor HA, Bond DS, Luke AK, Cardoso CC, Foster GD, Wing RR. Weight loss in Weight Watchers Online with and without an activity tracking device compared to control: A randomized trial. Obesity (Silver Spring). 2017 Jun;25(6):1014-1021. doi: 10.1002/oby.21846. Epub 2017 Apr 24. PMID 28437597